CLINICAL TRIAL: NCT04060550
Title: Investigate the Impact of Increased IgE on Innate Anti-herpes Simplex Virus 1 Responses in the Eczema Herpeticum Patients
Brief Title: Impact of Increased Immunoglobulin E to Anti-herpes Simplex Virus -1 Innate Immune Responses in Atopic Dermatitis Patients With Eczema Herpeticum
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML41620
Record Dates: First submitted 2019-08-07; First posted 2019-08-19 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Atopic Dermatitis With a History of Eczema Herpeticum; Atopic Dermatitis Without a History of Eczema Herpeticum; Health Controls Without Atopy
Keywords: Atopic dermatitis; Eczema herpeticum; Immunoglobulin E; Herpes simplex virus
MeSH Terms: conditions — Dermatitis, Atopic; Kaposi Varicelliform Eruption; Herpes Simplex | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood, monocytes purified from peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal controls: No history of skin disease and atopy
  Interventions: Biological: Xolair
- ADEH-: Atopic dermatitis without a history of eczema herpeticum
  Interventions: Biological: Xolair
- ADEH+: Atopic dermatitis with a history of eczema herpeticum
  Interventions: Biological: Xolair

INTERVENTIONS:
Biological: Xolair — This is in vitro mechanistic study. No drug will be given in vivo to patients.
  Other Names: omalizumab

SUMMARY:
This study investigates whether blood monocytes' surface bound- immunoglobulin E affects the innate immune responses against herpes simplex viruses in atopic dermatitis patients with eczema herpeticum.

DETAILED DESCRIPTION:
Some of atopic dermatitis patients (AD) have severe herpes simplex viral (HSV) infections, which could cause erosive skin lesions all over the body. This condition is termed as eczema herpeticum (ADEH+). Scientists have found that ADEH+ patients have significantly increased blood immunoglobulin (Ig) E compared to AD patients without eczema herpeticum and healthy people. Increased IgE in blood could bound to immune cells' surface, such as monocytes. Since monocytes serve as the first line defense to fight viral infection, their surface-bound IgE may interfere their anti-viral immune responses, and consequently results in more severe viral infections. The purpose of this study is to learn more about how increased IgE affect body's immune ability to fight herpes simplex viruses. This study includes three groups: AD patient without eczema herpeticum complication(ADEH-); AD patient with eczema herpeticum complication(ADEH+) and healthy controls. Study results will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-65 years old, age, sex and race match among non-atopic, ADEH- and ADEH+.
* Participant and/or parent guardian must be able to understand and provide informed consent, and fits in one of the following conditions:

  1. A history of AD with a history of eczema herpeticum, ADEH+, as diagnosed using the Atopic Dermatitis Research Network Standard Diagnostic Criteria.
  2. A history of AD without a history of eczema herpeticum, ADEH-, as diagnosed using Atopic Dermatitis Research Network Standard Diagnostic Criteria, and no first degree relatives with a history of EH.
  3. Non-atopic as diagnosed using Atopic Dermatitis Research Network Standard Diagnostic Criteria.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* Known or suspected immunosuppression
* Severe concomitant illness(es)
* Women of childbearing potential not using the contraception method(s) specified in this study (specify), as well as women who are breastfeeding
* Known sensitivity to study drug(s) or class of study drug(s)
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (specify as required)
* Use of any other investigational agent in the last 30 days

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: One of the following groups:
  1. A history of AD with a history of eczema herpeticum, ADEH+, as diagnosed using the Atopic Dermatitis Research Network Standard Diagnostic Criteria.
  2. A history of AD without a history of eczema herpeticum, ADEH-, as diagnosed using Atopic Dermatitis Research Network Standard Diagnostic Criteria, and no first degree relatives with a history of EH.
  3. Non-atopic as diagnosed using Atopic Dermatitis Research Network Standard Diagnostic Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Monocytes surface bound IgE quantities | One day
  Relative quantities of surface bound IgE

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States